CLINICAL TRIAL: NCT05995730
Title: Effect of Lavender Inhalation on Primary Dysmenorrhea
Brief Title: Effect of Lavender Inhalation on Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 16214662/050.01.04/130
Record Dates: First submitted 2023-06-13; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Lavender inhalation will be administered to this group.
  Interventions: Other: Lavender oil inhalation
- Placebo group (Placebo Comparator): Olive oil will be administered to the placebo group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lavender oil inhalation — Lavender inhalation will be administered to this group. Participants will be asked to drop three drops of lavender oil solution on a small piece of cotton on the 1st, 2nd, and 3rd days of their first menstrual bleeding after enrollment in the study, hold it 7-10 cm from their noses, and sniff for 5 minutes. Participants will be asked to apply this application immediately after the onset of dysmenorrhea pain on the first day of their menstruation and to continue regularly every 8 hours for the first three days of menstrual bleeding. Participants will be asked to apply this application in the same way in two consecutive menstrual cycles and the participants will be followed in this process.
  Arms: Experimental group
Other: Placebo — Olive oil will be administered to the placebo group. The application will be similar to the experimental group.
  Other Names: Olive oil
  Arms: Placebo group

SUMMARY:
This study was planned to determine the effect of lavender inhalation on primary dysmenorrhea and its symptoms.

DETAILED DESCRIPTION:
The research is a randomized controlled trial and an experimental research design will be used. The research will be carried out with two groups as experimental (lavender) and control (placebo) groups.

ELIGIBILITY:
Inclusion Criteria:

* Having primary dysmenorrhea (degrees II and III),
* Single,
* Who have never been pregnant before,
* Having a regular menstrual cycle
* Without any genital organ disorder (such as fibroids, fibroadenoma, endometriosis, metrorrhagia, ovarian cyst, pelvic inflammatory disease, chronic pelvic pain, other pelvic pathologies)
* Not using contraceptive method,
* Having a normal sense of smell
* People who can smell odors and are not allergic to odors will be included in the study.

Exclusion Criteria:

* Married,
* Having a disease that causes dysmenorrhea,
* Regularly using a pharmacological and non-pharmacological method to relieve
* Dysmenorrhea pain during the study,
* Having a previous or unconcluded pregnancy,
* Having a chronic disease (diabetes, endometriosis, uterine congenital anomalies, epilepsy, etc.),
* Using drugs that affect the menstrual cycle or dysmenorrhea,
* Persons who fill in the data collection form incompletely or not at all will not be included in the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Dysmenorrhea Symptom Assessment Form | to assess post-intervention change; It is applied on the 1st, 2nd and 3rd days of the menstrual cycle during 2 menstrual cycles.
  Form consists of questions about dysmenorrhea symptoms in the participants.As the score obtained from the form increases, the severity of the symptoms increases.
Numerical Pain Scale | to assess post-intervention change; It is applied on the 1st, 2nd and 3rd days of the menstrual cycle during 2 menstrual cycles.
  It will be applied to evaluate the level of dysmenorrhea pain. Participants will be asked to rate their pain level from 0 to 10. As the score increases, the level of pain increases

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Turkey (Türkiye)